CLINICAL TRIAL: NCT03496012
Title: A Randomised, Open Label, Outcomes-Assessor Masked, Prospective, Parallel Controlled Group, Phase 3 Clinical Trial of Retinal Gene Therapy for Choroideremia Using an Adeno-Associated Viral Vector (AAV2) Encoding Rab Escort Protein 1 (REP1)
Brief Title: Efficacy and Safety of BIIB111 for the Treatment of Choroideremia
Acronym: STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 273CH301; 2015-003958-41 (EudraCT Number: NightstaRx Ltd, a Biogen Company)
Record Dates: First submitted 2018-03-07; First posted 2018-04-12 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Choroideremia
Keywords: NightstaRx; NSR-REP1; Gene Therapy; AAV; REP1; Timrepigene Emparvovec
MeSH Terms: conditions — Choroideremia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BIIB111 High Dose (Experimental): Participants will receive a single administration of high dose BIIB111 in one eye through sub-retinal injection after vitrectomy.
  Interventions: Genetic: BIIB111
- BIIB111 Low Dose (Experimental): Participants will receive a single administration of low dose BIIB111 in one eye through sub-retinal injection after vitrectomy.
  Interventions: Genetic: BIIB111
- Untreated Control Group (No Intervention): Participants will receive no sham surgery or study medication.

INTERVENTIONS:
Genetic: BIIB111 — Administered as specified in the treatment arm.
  Other Names: AAV2-REP1
  Arms: BIIB111 High Dose; BIIB111 Low Dose

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of a single sub-retinal injection of BIIB111 in participants with choroideremia (CHM).

DETAILED DESCRIPTION:
This study was previously posted by NightstaRx Ltd. In October 2020, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Are willing and able to give informed consent for participation in the study.
* Have a documented genetically-confirmed diagnosis of CHM.
* Have active disease clinically visible within the macular region in the study eye.
* Have a BCVA of 34-73 ETDRS letters (equivalent to worse than or equal to 6/12 or 20/40 Snellen acuity, but better than or equal to 6/60 or 20/200 Snellen acuity) in the study eye.

Key Exclusion Criteria:

* Have a history of amblyopia in the eligible eye.
* Have had previous intraocular surgery performed in the study eye within 3 months of Visit 1.
* Have any other significant ocular or non-ocular disease/disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the results of the study, or the participant's ability to participate in the study.
* Have participated in another research study involving an investigational product in the past 12 weeks or received a gene/cell-based therapy at any time previously.
* Are unwilling to use barrier contraception methods, or abstain from sexual intercourse, for a period of 3 months, if treated with AAV2-REP1.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (18):
- United States (8):
  - Research Site, Los Angeles, California
  - Research Site, Miami, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Dallas, Texas
  - Research Site, Madison, Wisconsin
- Canada (2):
  - Research Site, Montreal
  - Research Site, Vancouver
- Research Site, Glostrup Municipality, Denmark
- Research Site, Helsinki, Finland
- Research Site, Montpellier, France
- Germany (2):
  - Research Site, Bonn
  - Research Site, Tübingen
- Research Site, Nijmegen, Netherlands
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Davis JL. The Blunt End: Surgical Challenges of Gene Therapy for Inherited Retinal Diseases. Am J Ophthalmol. 2018 Dec;196:xxv-xxix. doi: 10.1016/j.ajo.2018.08.038. Epub 2018 Sep 5. PMID 30194931

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the investigative sites in the United States, Germany, Finland, France, the United Kingdom, Canada, Netherlands, and Denmark from 11 December 2017 to 01 December 2020.
Pre-assignment Details: A total of 169 unique male participants with Choroideremia were randomized in the study (66 participants in Untreated Control Group; 34 participants in BIIB111 Low Dose group and 69 participants in BIIB111 High Dose group). Of which, 161 participants completed the study.
Groups:
- Untreated Control Group: Participants received no sham surgery or study medication to allow for a controlled comparison.
- BIIB111 Low Dose: Followed by vitrectomy and retinal detachment in the study eye, participants received a single administration of low dose (1 × 10^10 genome particle [gp]) BIIB111 (timrepigene emparvovec) as a sub-retinal injection on Day 0 (surgery day).
- BIIB111 High Dose: Followed by vitrectomy and retinal detachment in the study eye, participants received a single administration of high dose (1 × 10^11 gp) BIIB111 (timrepigene emparvovec) as a sub-retinal injection on Day 0 (surgery day).
Period: Overall Study
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Started | 66 | 34 | 69
Completed | 62 | 34 | 65
Not Completed | 4 | 0 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Reason Not Specified | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who either received study treatment (BIIB111) or a post-randomization study visit (control group).
Groups:
- BIIB111 Low Dose: Followed by vitrectomy and retinal detachment in the study eye, participants received a single administration of low dose (1 × 10^10 gp) BIIB111 (timrepigene emparvovec) as a sub-retinal injection on Day 0 (surgery day).
- Total: Total of all reporting groups
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose | Total
Number analyzed (Participants) | 65 | 34 | 65 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (13.73) | 49.8 (12.62) | 47.5 (12.91) | 48.7 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 65 | 34 | 65 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4 | 8
  Not Hispanic or Latino | 51 | 26 | 54 | 131
  Unknown or Not Reported | 11 | 7 | 7 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 0 | 1 | 1
  Race: American Indian or Alaska Native | 1 | 0 | 0 | 1
  Race: Black or African American | 1 | 0 | 0 | 1
  Race: White | 55 | 30 | 59 | 144
  Race: Other | 1 | 0 | 0 | 1
  Race: Not Reported | 7 | 4 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥15 -Letter Improvement From Baseline in Best Corrected Visual Acuity (BCVA) at Month 12 as Measured by the Early Treatment of Diabetic Retinopathy Study (ETDRS) Chart
Description: BCVA was assessed for both eyes using the ETDRS visual acuity (VA) chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of participants with a ≥15 -letter improvement from baseline in BCVA at Month 12 was reported for both eyes.
Time Frame: Month 12
Population: Intent-to-treat (ITT) population included all randomized participants who received the study treatment (or the phone call for those in the untreated control group) and had at least one post-treatment BCVA measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 62 | 34 | 65
percentage of participants
  Study Eye | 0 [0 to 5.8] | 2.9 [0.1 to 15.3] | 4.6 [1.0 to 12.9]
  Fellow Eye | 0 [0 to 5.8] | 0 [0 to 10.3] | 3.1 [0.4 to 10.7]
Statistical Analysis 1: Comparison: Untreated Control Group vs BIIB111 Low Dose; Test type: Superiority; p = 0.354, Fisher's Exact; Difference in Proportions = 2.9, 95% CI 2-sided [-3.1 to 15]
Statistical Analysis 2: Comparison: Untreated Control Group vs BIIB111 High Dose; Test type: Superiority; p = 0.245, Fisher's Exact; Difference in proportions = 4.6, 95% CI 2-sided [-1.4 to 12.8]

2. Secondary Outcome: Change From Baseline in BCVA at Month 12 Reported as Letters Measured by the ETDRS Chart in Study Eye
Description: BCVA was assessed for study eye using the ETDRS VA chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. BCVA was reported as number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). An increase in the number of letters read correctly means that vision has improved. Here negative values indicate decline in BCVA.
Time Frame: Baseline, Month 12
Population: ITT population included all randomized participants who received the study treatment (or the phone call for those in the untreated control group) and had at least one post-treatment BCVA measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: letters
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 62 | 34 | 65
letters | -2.3 [-5.31 to 0.61] | -1.5 [-5.47 to 2.50] | -0.3 [-3.18 to 2.64]

3. Secondary Outcome: Percentage of Participants With a ≥10 -Letter Improvement From Baseline in BCVA at Month 12 Measured by the ETDRS Chart
Description: BCVA was assessed for both eyes using the ETDRS VA chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of participants with a ≥10 -letter improvement from baseline in BCVA at Month 12 was reported for both eyes.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 62 | 34 | 65
percentage of participants
  Study Eye | 1.6 [0.0 to 8.7] | 17.6 [6.8 to 34.5] | 13.8 [6.5 to 24.7]
  Fellow Eye | 0 [0.0 to 5.8] | 8.8 [1.9 to 23.7] | 6.2 [1.7 to 15.0]
Statistical Analysis 1: Comparison: Untreated Control Group vs BIIB111 Low Dose; Test type: Superiority; Difference in proportions = 16, 95% CI 2-sided [5.3 to 32.2]
Statistical Analysis 2: Comparison: Untreated Control Group vs BIIB111 High Dose; Test type: Superiority; Difference in proportions = 12.2, 95% CI 2-sided [3.5 to 23]

4. Secondary Outcome: Percentage of Participants With No Decrease From Baseline in BCVA or a Decrease From Baseline in BCVA of <5 ETDRS Letters at Month 12 Measured by the EDRS Chart
Description: BCVA was assessed for both eyes using the ETDRS VA chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). Percentage of participants with no decrease or a decrease of <5 letters from baseline in BCVA at Month 12 was reported for both eyes.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 62 | 34 | 65
percentage of participants
  Study Eye | 67.7 [54.7 to 79.1] | 70.6 [52.5 to 84.9] | 83.1 [71.7 to 91.2]
  Fellow Eye | 75.8 [63.3 to 85.8] | 85.3 [68.9 to 95.0] | 90.8 [81.0 to 96.5]
Statistical Analysis 1: Comparison: Untreated Control Group vs BIIB111 Low Dose; Test type: Superiority; Difference in proportions = 2.8, 95% CI 2-sided [-17.2 to 21]
Statistical Analysis 2: Comparison: Untreated Control Group vs BIIB111 High Dose; Test type: Superiority; Difference in proportions = 15.3, 95% CI 2-sided [0.3 to 30.1]

5. Secondary Outcome: Change From Baseline in BCVA at Months 4 and 8 Reported as Letters Measured by the ETDRS Chart
Description: BCVA was assessed for both eyes using the ETDRS VA chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. BCVA was reported as number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters) in both the study and fellow eyes. The lower the number of letters read correctly on the eye chart, the worse the vision (or VA). An increase in the number of letters read correctly means that vision has improved. Here negative values indicate decline in BCVA.
Time Frame: Baseline, Months 4 and 8
Population: ITT population included all randomized participants who received the study treatment (or the phone call for those in the untreated control group) and had at least one post-treatment BCVA measurement. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 61 | 34 | 65
letters
  Change From Baseline at Month 4: Study Eye | 0.2 (4.34) | -0.4 (14.16) | 0.6 (11.11)
  Change From Baseline at Month 4: Fellow Eye: number analyzed (Participants) | 61 | 34 | 64
  Change From Baseline at Month 4: Fellow Eye | -1.1 (8.45) | 0.9 (6.67) | 2.0 (6.63)
  Change From Baseline at Month 8: Study Eye | -0.8 (4.93) | -1.1 (13.13) | 0.1 (11.71)
  Change From Baseline at Month 8: Fellow Eye: number analyzed (Participants) | 61 | 34 | 64
  Change From Baseline at Month 8: Fellow Eye | -0.4 (8.31) | 1.9 (7.06) | 1.6 (5.91)

6. Secondary Outcome: Change From Baseline in Total Area of Preserved Autofluorescence (AF) at Month 12 in Study Eye
Description: Fundus AF was used to assess change in total area of preserved AF. Areas of preserved AF were identified as well-demarcated regions of relative hyper AF compared with the background areas of surrounding atrophy. A negative change from baseline indicate decline in total area of preserved AF.
Time Frame: Baseline, Month 12
Population: ITT population included all randomized participants who received the study treatment (or the phone call for those in the untreated control group) and had at least one post-treatment BCVA measurement. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Least Squares Mean (Standard Error); unit: square millimeters (mm^2)
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 57 | 34 | 63
square millimeters (mm^2) | -0.3872 (0.0389) | -0.5413 (0.0501) | -0.5136 (0.0371)

7. Secondary Outcome: Change From Baseline in Distance From Foveal Center to Nearest Border of Preserved AF at Month 12 in Study Eye
Description: Fundus AF was used to assess change in distance from foveal center (FC) to nearest border of preserved AF. A negative change from baseline indicate decline in distance from FC to nearest border of AF.
Time Frame: Baseline, Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: micrometers (µm)
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 57 | 34 | 63
micrometers (µm) | 21.7796 (9.6234) | 23.6171 (12.3765) | 21.1660 (9.1863)

8. Secondary Outcome: Change From Baseline in the Foveal Subfield Thickness Using Spectral Domain Optical Coherence Tomography (SD-OCT) at Month 12 in Study Eye
Description: SD-OCT was used to assess change in foveal subfield thickness. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates decline in foveal subfield thickness.
Time Frame: Baseline, Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: µm
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 61 | 34 | 64
µm | -6.3152 (2.7779) | -19.8654 (3.6998) | -15.7993 (2.7233)

9. Secondary Outcome: Change From Baseline in the Total Macular Volume Using SD-OCT at Month 12 in Study Eye
Description: SD-OCT was used to assess change in total macular volume. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates decline in total macular volume.
Time Frame: Baseline, Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: cubic millimeters (mm^3)
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 61 | 34 | 64
cubic millimeters (mm^3) | -0.0895 (0.0485) | -0.2876 (0.0646) | -0.2088 (0.0476)

10. Secondary Outcome: Change From Baseline in the Central Horizontal Ellipsoid Width Using SD-OCT at Month 12 in Study Eye
Description: SD-OCT was used to assess change in central horizontal ellipsoid width. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates decline in central horizontal ellipsoid width.
Time Frame: Baseline, Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: µm
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 59 | 32 | 60
µm | -81.9178 (20.6192) | -116.3811 (27.8213) | -170.7214 (20.4062)

11. Secondary Outcome: Change From Baseline in the Central Ellipsoid Area Using SD-OCT at Month 12 in Study Eye
Description: SD-OCT was used to assess change in central ellipsoid area. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates decline in central ellipsoid area.
Time Frame: Baseline, Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 37 | 18 | 44
mm^2 | -0.2382 (0.0364) | -0.4229 (0.0527) | -0.3440 (0.0332)

12. Secondary Outcome: Change From Baseline in the Choroidal Thickness Using SD-OCT at Month 12 in Study Eye
Description: SD-OCT was used to assess change in choroidal thickness. The measurements were taken after dilation of the participant's pupil. A negative change from baseline indicates decline in choroidal thickness.
Time Frame: Baseline, Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: µm
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 61 | 34 | 64
µm | -5.4897 (2.1873) | -7.9579 (2.9207) | -4.6371 (2.1446)

13. Secondary Outcome: Change From Baseline in the Mean Retinal Sensitivity Using Microperimetry at Month 12 in Study Eye
Description: Microperimetry was conducted to assess change in mean retinal sensitivity within the macula. Retinal mean sensitivity to light was measured in decibels (dBs) in multiple spots across the central and peripheral retina (entire visual field). Higher numbers (dBs) indicate higher retinal sensitivity. A negative change from baseline indicates decline in retinal sensitivity.
Time Frame: Baseline, Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: dBs
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 58 | 34 | 61
dBs | -0.3443 (0.1134) | -0.2965 (0.1478) | -0.5015 (0.1112)

14. Secondary Outcome: Change From Baseline in the Bivariate Contour Ellipse Area 63% Using Microperimetry at Month 12 in Study Eye
Description: Microperimetry was conducted to assess change in bivariate contour ellipse area 63%. A negative change from baseline indicates decline in bivariate contour ellipse area 63%.
Time Frame: Baseline, Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: square degrees (deg^2)
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 58 | 34 | 61
square degrees (deg^2) | -3.2161 (1.2623) | -3.3771 (1.6405) | -2.5555 (1.2403)

15. Secondary Outcome: Change From Baseline in the Bivariate Contour Ellipse Area 95% Using Microperimetry at Month 12 in Study Eye
Description: Microperimetry was conducted to assess change in bivariate contour ellipse area 95%. A negative change from baseline indicates decline in bivariate contour ellipse area 95%.
Time Frame: Baseline, Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: deg^2
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 58 | 34 | 61
deg^2 | -10.1986 (4.1004) | -14.6926 (5.3134) | -11.6863 (4.0207)

16. Secondary Outcome: Change From Baseline in Contrast Sensitivity Score at Month 12 in Study Eye
Description: Change in contrast sensitivity was assessed by Pelli-Robson chart which uses a single large letter size (20/60 optotype), with contrast varying across groups of letters (6 per line), whose contrast varies from high to low. Participants read letters, starting with highest contrast, until they are unable to read 2 or 3 letters in a single group. Each group had three letters of the same contrast level, so there were three trials per contrast level. Score is assigned based on contrast of last group in which 2 or 3 letters were correctly read. Score is a measure of participant's log contrast sensitivity ranging from 0 (no letters read) to 2.25 (all letters read). Total CS score=[(total letters correct-3) x 0.05]. A negative change from baseline indicates worsening in contrast sensitivity score.
Time Frame: Baseline, Month 12
Population: ITT population included all randomized participants who received study treatment (phone call for untreated control group) and had at least 1 post-treatment BCVA measurement. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 60 | 34 | 65
score on a scale | -0.0595 (0.0315) | -0.0130 (0.0417) | -0.0386 (0.0304)

17. Secondary Outcome: Change From Baseline in Colour Vision Total Error Score at Month 12 in Study Eye
Description: Colour vision total error scores were assessed by the Farnsworth Munsell 100 Hue Sort Test. Farnsworth Munsell 100 Hue Test requires placing 100 colour palettes in the correct order based upon colour hue. Scores are determined by the frequency and severity of any displacement in the correct order. One error equates to one misplaced hue, by one step or position. An error score of 0 indicates no errors in ordering the hues while error score greater than 500 indicates virtually no color discrimination. A Total Error Score of 0 to 128 could be seen in a normal population.
Time Frame: Baseline, Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 51 | 28 | 51
score on a scale | 35.0003 (23.5973) | 43.5915 (31.7720) | 54.3777 (24.0358)

18. Secondary Outcome: Change From Baseline in Reading Speed Test at Month 12 in Study Eye
Description: The reading speed (words per minute) was calculated using the following formula: [number of words in the text - number of misread words] / reading time x 60. The number of misread words and reading time is collected. A negative change from baseline indicates decline in reading speed.
Time Frame: Baseline, Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: words per minute
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 23 | 12 | 27
words per minute | -149.5590 (10.9857) | -122.1333 (14.3276) | -127.4706 (9.9110)

19. Secondary Outcome: Change From Baseline in the 25-Item Visual Function Questionnaire (VFQ-25) Composite Scores at Month 12 in Study Eye
Description: VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. A score of 0 represents the worst outcome and 100 represents the best outcome. A negative change from baseline indicates decline in VFQ-25 score.
Time Frame: Baseline, Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
Number analyzed (Participants) | 58 | 34 | 63
score on a scale | -2.6971 (1.2786) | 1.7236 (1.6624) | 0.7964 (1.2308)

ADVERSE EVENTS:
Time Frame: From signing of informed consent through end of study (up to 12 months)
Description: Safety population included all randomized participants who either received study treatment (BIIB111) or a post-randomization study visit (control group).
Arm/Group | Untreated Control Group | BIIB111 Low Dose | BIIB111 High Dose
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/34 | 0/65
Serious Adverse Events (participants affected / at risk) | 10/65 | 9/34 | 11/65
Other Adverse Events (participants affected / at risk) | 9/65 | 30/34 | 54/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Untreated Control Group (N=65) | BIIB111 Low Dose (N=34) | BIIB111 High Dose (N=65)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Heterophoria (Eye disorders) | 0 | 0 | 1
Macular hole (Eye disorders) | 1 | 0 | 1
Noninfective retinitis (Eye disorders) | 0 | 0 | 1
Retinal artery embolism (Eye disorders) | 1 | 0 | 0
Retinal vascular occlusion (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 8 | 5 | 5
Visual impairment (Eye disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Covid-19 pneumonia (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Untreated Control Group (N=65) | BIIB111 Low Dose (N=34) | BIIB111 High Dose (N=65)
Intraocular pressure increased (Investigations) | 0 | 1 | 6
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Ocular procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 5
Headache (Nervous system disorders) | 0 | 3 | 7
Anterior chamber cell (Eye disorders) | 0 | 14 | 24
Anterior chamber flare (Eye disorders) | 0 | 2 | 4
Cataract (Eye disorders) | 3 | 3 | 9
Blepharitis (Eye disorders) | 0 | 2 | 1
Cataract subcapsular (Eye disorders) | 0 | 4 | 4
Conjunctival haemorrhage (Eye disorders) | 0 | 13 | 26
Conjunctival hyperaemia (Eye disorders) | 0 | 4 | 7
Eye irritation (Eye disorders) | 0 | 5 | 8
Eye pain (Eye disorders) | 0 | 6 | 11
Glare (Eye disorders) | 0 | 2 | 1
Foreign body sensation in eyes (Eye disorders) | 0 | 3 | 9
Low luminance best-corrected visual acuity decreased (Eye disorders) | 0 | 2 | 7
Ocular hyperaemia (Eye disorders) | 0 | 4 | 7
Ocular discomfort (Eye disorders) | 0 | 0 | 6
Retinal haemorrhage (Eye disorders) | 1 | 3 | 2
Vision blurred (Eye disorders) | 0 | 3 | 1
Vitritis (Eye disorders) | 0 | 10 | 16
Vitreal cells (Eye disorders) | 0 | 3 | 4
Initial insomnia (Psychiatric disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Impetigo (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 4 | 3 | 6
Pneumonia (Infections and infestations) | 0 | 2 | 2
Sinusitis (Infections and infestations) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT03496012/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT03496012/SAP_001.pdf